CLINICAL TRIAL: NCT00917033
Title: Orotracheal Intubation of Morbidly Obese Patients. A Randomised Controlled Trial Comparing the GlideScope Videolaryngoscope to the Macintosh Direct Laryngoscope.
Brief Title: Tracheal Intubation of Morbidly Obese Patients. GlideScope Versus Direct Laryngoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Mr. Lasse Hoegh Andersen, M.D., Department of Anaesthesia, Glostrup University Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LHA GS 01
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Intubation, Endotracheal; Anesthesia, General; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GlideScope (Experimental): Orotracheal intubation using the GlideScope videolaryngoscope
  Interventions: Device: GlideScope
- Macintosh (Active Comparator): Orotracheal intubation using the Macintosh direct laryngoscope
  Interventions: Device: Macintosh direct laryngoscope

INTERVENTIONS:
Device: GlideScope — Orotracheal intubation
  Arms: GlideScope
Device: Macintosh direct laryngoscope — Orotracheal intubation
  Arms: Macintosh

SUMMARY:
The purpose of this study is to examine whether orotracheal intubation in morbidly obese patients is faster, gentler and safer using the GlideScope videolaryngoscope than with the Macintosh direct laryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* Approved for elective bariatric surgery at Glostrup University Hospital, Copenhagen.
* Body Mass Index at least 35 kg/m2
* Written informed consent to participate

Exclusion Criteria:

* Mental illness
* Abuse of alcohol or other substances
* Previous difficult tracheal intubation
* Considered non-eligible for safety-reasons by the anesthetist in charge

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2008-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Time to intubate | Measured during intubation (seconds)

SECONDARY OUTCOMES:
Number of intubation attempts | Measured during intubation (seconds)
Lowest arterial oxygen saturation during intubation | Measured during intubation (seconds)
Subjective difficulty of intubation | Measured during intubation (seconds)
Cormack-Lehane Score | Measured during intubation (seconds)
Airway mucosal trauma | Measured during intubation (seconds)
Dental injury | Measured during intubation (seconds)
Post-procedure sore throat | One hour post-operative
Post-procedure hoarseness of voice | One hour post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Lasse H Andersen, MD, Principal Investigator — Glostrup University Hospital
Locations (1):
- Department of Anesthesia, Glostrup University Hospital, Copenhagen, Glostrup, Denmark